CLINICAL TRIAL: NCT01394926
Title: A Multi-Center, Open-Label, Dose-Finding, Feasibility Study of Optison in Contrast Enhanced U/S for the Detection of Carotid Artery Disease
Brief Title: Dose-Finding, Feasibility Study of Optison in Contrast Enhanced U/S for the Detection of Carotid Artery Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Subject Recruitment
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-191-001
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Carotid Artery Disease
Keywords: CE-U/S - Contrast-Enhanced U/S; U/S - Ultrasound; Assess effectiveness
MeSH Terms: conditions — Carotid Artery Diseases | interventions — FS 069

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm Number 1 (Experimental)
  Interventions: Drug: Optison

INTERVENTIONS:
Drug: Optison — Optison is a sterile non-pyrogenic suspension of perflutren for IV administration.
  Other Names: Perflutren Protein-Type A Microspheres Injectable Suspension, USP

SUMMARY:
The purpose of this study is to find the optimal dose from 3 different dose levels - 0.15 mL, 0.5 mL and 1.5 mL of Optison in assessing the presence of disease of the carotid arteries when comparing pre-contrast to post-contrast ultrasound (U/S) by dose group.

ELIGIBILITY:
Inclusion Criteria:

* The subject is is greater than or equal to 18 years of age.
* The subjects has highly suspected or established carotid artery disease.
* The subject has undergone or been referred for either unilateral or bilateral intra-arterial X-ray carotid angiography for the determination of subject management (within 30 days before or after the U/S procedure).
* The subject has non-diagnostic U/S of the carotids as defined by institutional standards.

Exclusion Criteria:

* The subject presents any clinically active, serious, life-threatening disease, with a life expectancy of less than 1 month or where study participation may compromise the management of the subject or other reason that in the judgment of the investigator makes the subject unsuitable for participation in the study.
* The subject has a history of acute occlusion requiring medical intervention of any artery (including aorta) within 6 months of consent.
* The subject has a known or suspected hypersensitivity to any of the components of Optison, blood, blood products, or albumin.
* The subject has right to left, bi-directional or transient right to left cardiac shunts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Perrone, M.D., Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 Subjects enrolled in study. 21 subjects completed this study. 0 subjects did not complete the study.
Period: Overall Study
Arm/Group | Optison
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Optison
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (9.40)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Finding the Optimal Dose of Optison From 3 Different Dose Levels; 0.15mL, 0.5mL, and 1.5mL.
Description: Assessing the presence of disease of the carotid arteries when comparing pre-contrast to post-contrast ultrasound (U/S) by dose group. Using the optimal dose from 3 different dose levels - 0.15 mL, 0.5 mL and 1.5 mL of Optison.
Time Frame: Up to 10 minutes post contrast administration.
Population: Due to difficulty enrolling subjects in all three dose levels of Optison, this study was stopped prematurely. No efficacy analyses were performed.
Groups:
- Dose Level 1: Injection of 0.15mL Optison at Time 0.: Dose Level 1 given as an Injection of 0.15mL of Optison at time 0.
- Dose Level 2: 0.5mL of Optsion at Time 6.5 Minutes: Dose Level 2: Inj. of 0.5mL Optsion at time 6.5 minutes post dose level 1.
- Dose Level 3: 1.5mL Optison 8 Minutes: Dose Level 3: Injection of 1.5mL of Optison 8 minutes post level 2.
Arm/Group | Dose Level 1: Injection of 0.15mL Optison at Time 0. | Dose Level 2: 0.5mL of Optsion at Time 6.5 Minutes | Dose Level 3: 1.5mL Optison 8 Minutes
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Detecting the Presence of Greater Than or Equal to 50% Stenosis and Greater Than or Equal to 75% Stenosis in the Carotid Arteries When Comparing Pre-contrast to Post-contrast Ultrasound by Dose Group.
Description: Detecting the presence of greater than or equal to 50% stenosis and greater than or equal to 75% stenosis in the carotid arteries when comparing pre contrast to post-contrast U/S by dose group.Using the 3 different dose levels of 0.15 mL, 0.5 mL and 1.5 mL of Optison.
Time Frame: Up to 10 minutes post contrast administration.
Population: Due to difficulty enrolling subjects in all three dose levels of Optison , this study was stopped prematurely. No efficacy analyses were performed.
Groups:
- Dose Level 1: Injection of 0.15mL Optison at Time 0.: Dose Level 1: Injection of 0.15mL Optison at time 0.
- Dose Level 2: 0.5mL Optison at Time 6.5 Minutes: Dose Level 2: Injection given of 0.5mL of Optison at 6.5 minutes post dose level 1.
- Dose Level 3: 1.5mL Optison 8 Minutes: Dose Level 3: Injection of 1.5mL of Optison 8 minutes post dose level 2.
Arm/Group | Dose Level 1: Injection of 0.15mL Optison at Time 0. | Dose Level 2: 0.5mL Optison at Time 6.5 Minutes | Dose Level 3: 1.5mL Optison 8 Minutes
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Optison
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 2/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optison (N=21)
Dysgeusia (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No